CLINICAL TRIAL: NCT00828607
Title: Characterization of Liver Masses With Contrast Enhanced Ultrasound (CEUS): A Comparison With Standard Institutional Contrast Enhanced CT (CECT) or MR Scan (CEMRI)
Brief Title: Contrast Enhanced (CE) Ultrasound and CE Computed Tomography or CE Magnetic Resonance Imaging in Liver Masses
Status: Completed | Type: Observational
Sponsor: Foothills Medical Centre (Other)
Collaborators: Vancouver General Hospital (Other); London Health Sciences Centre (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Stephanie R Wilson, MD, Clinical Professor University of Calgary, Foothills Medical Centre
Other Study IDs: (Ethics ID: 21295)
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Liver Tumors
Keywords: Contrast Enhanced Ultrasound (CEUS); Liver tumors; Hepatocellular carcinoma; Hemangioma; Focal Nodular Hyperplasia; Hepatic metastases
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hemangioma; Focal Nodular Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- liver mass: The group will comprise any patients with an unknown liver mass at the time of diagnostic imaging.

SUMMARY:
This comparison study is performed to show equivalence of CEUS with CECT or CEMR to diagnose noninvasively focal liver masses. This is a multi-center prospective cohort study of 250 subjects, which will be performed at four institutions in Canada. Subjects with a focal liver mass, measuring at least 2.5 centimeters in maximal diameter, will undergo a conventional baseline sonogram followed by a contrast enhanced ultrasound (CEUS). CEUS will be performed on standard ultrasound scanners with contrast specific imaging capability. The contrast agent used is Definity (Lantheus Medical Imaging, Billerica,MA) All subjects will have either a dedicated hepatic contrast enhanced CT or MR scan within 60 days of the CEUS as per the standard of care in the institution. Anonymized image files from all imaging will be shown independently to two readers, blinded to all clinical and demographic data, who will predict malignancy and diagnosis.

DETAILED DESCRIPTION:
This comparison study is performed to show equivalence of CEUS with CECT or CEMR to diagnose noninvasively focal liver masses. This is a multi-center prospective cohort study of 250 subjects, which will be performed at four institutions in Canada. Subjects with a focal liver mass, measuring at least 2.5 centimeters in maximal diameter, will undergo a conventional baseline sonogram followed by a contrast enhanced ultrasound (CEUS). CEUS will be performed on standard ultrasound scanners with contrast specific imaging capability. The contrast agent used is Definity (Lantheus Medical Imaging, Billerica,MA) All subjects will have either a dedicated hepatic contrast enhanced CT or MR scan within 60 days of the CEUS as per the standard of care in the institution. Anonymized image files from all imaging will be shown independently to two readers, blinded to all clinical and demographic data, who will predict malignancy and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* An incidental liver mass amenable to US evaluation
* Undiagnosed liver mass
* Mass threshold size is 2.5 cm
* Source of subjects:

  * Liver mass found on conventional institutional US
  * Liver mass detected on CT and MRI that remain uncategorized
  * Referral of patient with a liver mass following detection in outside institution.
* Confirmatory CT or MRI performed within 60 days of initial scan according to the institutional protocols

Exclusion Criteria:

* Any known pre existing mass
* Pregnancy
* Severe or unstable cardiac disease, including angina, congestive heart failure, or arrhythmias
* Severe COPD
* Pulmonary hypertension
* Bidirectional shunts
* Transient right to left shunts
* Known hypersensitivity to Definity or any of its components

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with an unknown liver mass
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2009-01; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Malignancy of the liver mass, as determined on US, on CEUS, and on CECT or CEMRI. | 6-9 months

SECONDARY OUTCOMES:
Diagnosis of the liver mass, as determined on US, on CEUS, and on CECT or CEMRI. | 6-9 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie R Wilson, MD, Principal Investigator — Foothills Medical Centre
Locations (4):
- Canada (4):
  - Vancouver General Hospital, Vancouver, British Columbia
  - London Health Sciences Centre, University Hospital, London, Ontario
  - Sunnybrook Medical centre, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal, Hôpital Saint-Luc, Montreal, Quebec